CLINICAL TRIAL: NCT04378361
Title: CONFORM-TAD- A Post-market Clinical Follow-up Study in Patients With Complicated Acute, Subacute or Chronic Type B Aortic Dissection With Double Lumen Treated With the E-nya Thoracic Stent Graft System
Brief Title: A Study in Patients With Complicated Type B Aortic Dissection Treated With the E-nya Thoracic Stent Graft
Acronym: CONFORM-TAD
Status: Withdrawn | Type: Observational
Why Stopped: Expiry of CE mark.
Sponsor: JOTEC GmbH (Industry)
Collaborators: MedPass International (Industry)
Responsible Party: Sponsor
Other Study IDs: CONFORM-TAD
Record Dates: First submitted 2020-05-03; First posted 2020-05-07 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Vascular Diseases
Keywords: Descending; Aorta; Dissection; Complicated
MeSH Terms: conditions — Vascular Diseases | interventions — Endovascular Aneurysm Repair

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: endovascular repair — Endovascular repair of complicated acute, subacute or chronic type B aortic dissection with double lumen

SUMMARY:
The CONFORM-TAD post-market clinical follow-up study is undertakento evaluate the prevention of death related to the treatment of a complicated acute, subacute or chronic type B aortic dissection with the E-nya Thoracic Stent Graft System. The secondary objective is to evaluate safety and clinical performance of the device.

DETAILED DESCRIPTION:
In this study, patients who receive an E-nya Thoracic Stent Graft for the treatment of a complicated acute, subacute or chronic type B aortic dissection will be observed. The E-nya Thoracic Stent Graft will be implanted in accordance with the instructions for use of the E-nya Thoracic Stent Graft System and at the discretion of the treating physician.

Participating physicians will be asked to provide their observations collected during routine standard of care for patients he/she had decided to treat with the E-nya Thoracic Stent Graft System. Informed consent of the patients will be obtained to allow the use of their clinical records for the purpose of this observational study before data are being collected.

The period of data collection for each patient will be approximately 60 months from the intervention. Source document verification will be performed on 100% of patients; data from all visits will be reviewed and verified against existing source documents. Complete DICOM image files of the CT scans will be sent to the CoreLab for independent evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 85 years
* Complicated acute, subacute or chronic type B aortic dissection with evidence of at least one of the following:

  * Malperfusion (visceral, renal, spinal cord and/or lower limb ischemia)
  * Three of the following risk factors in acute or subacute dissections

    * Young patient
    * Primary entry tear > 10 mm
    * Early aortic expansion > 5 mm within 6 months
    * Total aortic diameter > 40 mm
    * False lumen diameter > 20 mm
    * Partially thrombosed false lumen
  * Total diameter > 50 mm in case of chronic dissections
* Patient is hemodynamically stable (stable blood pressure and heart rate, no shock)
* Planned proximal and distal landing zone of the E-nya Thoracic Stent Graft component(s) in the native aorta
* Landing zone of the proximal edge of the fabric distal to the left carotid artery
* Landing zone of the distal edge of the fabric proximal to the celiac trunk
* Proximal landing zone diameter between 20 and 44 mm
* Centerline distance from the distal edge of the left carotid artery to the start of the most proximal tear ≥ 20 mm
* Thoracic aortic lesion confirmed by thin sliced (≤ 1 mm) CTA with optional three-dimensional reconstruction obtained within 3 months prior to the implant procedure
* Patient is able and willing to undergo follow-up imaging and examinations prior to discharge from the hospital, at 30 days and 12 months, and annually thereafter until 5 years follow-up
* Patient understands and has signed the Informed Consent Form prior to intervention whenever possible or after the intervention in case the patient's status does not allow consent to be obtained prior to intervention

Exclusion Criteria:

* Female of child bearing potential, breast feeding
* Access vessels not suitable for endovascular treatment
* Significant circular thrombi or calcification in proximal or distal landing zones
* Genetic connective tissue diseases (e.g. Marfan Syndrome or Ehlers-Danlos Syndrome)
* Allergies against materials necessary for endovascular repair (e.g. contrast media, heparin, materials of the stent graft)
* Systemic or local infections
* eGFR < 45 ml/min/1.73m2 before the intervention
* Myocardial infarction or cerebrovascular accident < 3 months
* Patient has specified disease of the thoracic aorta which is not included in the registry, for example: intramural hematoma, penetrating aortic ulcer, traumatic injury or transection, (contained) aortic rupture (hemorrhage outside of aorta)
* Patients who are planned to be treated with a chimney in the left subclavian artery
* Patients who are planned to be treated with the Petticoat concept
* Previous stent and/or stent graft or previous surgical repair of descending thoracic aorta
* Patient had or planned to have a major surgical or interventional procedure within 30 days before or 30 days after the planned implantation of the E-nya Stent Graft System(s). This exclusion does not include planned procedures that are needed for the safe and effective placement of the stent graft (ie, carotid/subclavian transposition, carotid/subclavian bypass procedure)
* Other medical condition that may cause the patient to be non-compliant with the protocol, confound the results, or is associated with a limited life expectancy (i.e. heart failure, active malignancy (progressive, stable or partial remission))
* Simultaneously participating in another clinical trial
* NYHA class IV

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female patients with complicated acute, subacute or chronic type B aortic dissection and who are eligible for treatment with a thoracic stent graft according to the instructions for use for the E-nya Thoracic Stent Graft System and scheduled for implantation of the E-nya Stent Graft System at their physician's discretion in accordance with the listed inclusion / exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-05-25 (Actual); Primary Completion 2024-07-24 (Actual); Study Completion 2024-07-24 (Actual)

PRIMARY OUTCOMES:
Mortality | 30-day
  Rate of all-cause mortality

SECONDARY OUTCOMES:
Mortality | 24 hours
  Rate of all-cause mortality
Mortality | 12, 24, 36, 60 months
  Rate of all-cause mortality
Dissection related mortality | 30-day, 12, 24, 36, 60 months
  Rate of dissection related mortality
Primary technical success | 24 hours
  Primary technical success related to the E-nya Thoracic Stent Graft System combines the following criteria:
  * It is related to periprocedural events that occur from the initiation of the procedure and extend through the first 24-hours postoperative period
  * Defined on an intent-to-treat basis
  * Successful access to the arterial system using a remote site (ie, the femoral, external iliac, common iliac, abdominal aorta, or brachiocephalic arteries with or without use of a temporary or permanent prosthetic conduit to access these arteries)
  * Successful deployment of the endoluminal graft at the intended location
  * Coverage of the primary entry tear
  * Absence of reintervention, surgical conversion to open repair or death ≤24 h
  * Patent endoluminal graft
Technical success | 24 hours
  Technical success is achieved in case all above mentioned criteria are fulfilled however, a reintervention was performed.
Primary clinical success | prior to discharge/30-day, 12, 24, 36, and 60 months
  Primary clinical success related to the E-nya Thoracic Stent Graft combines the following criteria:
  * Clinical success should be reported on an intent-to-treat basis
  * Initially required successful deployment of the E-nya Thoracic Stent Graft at the intended location without any
    * Death as a result of the pathology that was treated
    * Conversion to open repair
    * Reintervention
    * E-nya Thoracic Stent Graft infection
    * E-nya Thoracic Stent Graft infolding
    * Causing a new thoracic aortic pathology as a result of the intervention (e.g. pseudoaneurysm, dissection, intramural hematoma)
Clinical success | prior to discharge/30-day, 12, 24, 36, and 60 months
  Clinical success is achieved in case all above mentioned criteria are fulfilled however, a reintervention was performed.
Major Adverse Events (MAE) | 30-day, 12, 24, 36, 60 months
  • Rate of patients with major adverse event(s) (death, aneurysm rupture , conversion to open surgical repair, retrograde type A dissection, stent graft induced new entry tear requiring intervention, new myocardial infarction requiring intervention (percutaneous transluminal coronary angioplasty, bypass), new disabling stroke, new permanent paraplegia, new permanent paraparesis, new chronic renal insufficiency/renal failure requiring dialysis, bowel resection, > 72 hours artificial respiratory assistance, device induced trauma requiring intervention) product-related, procedure-related, dissection-related)
Conversion to open surgical repair | 24 hours, 30-day, 12, 24, 36, 60 months
  Rate of patients with conversion to open surgical repair
Size of true lumen | prior to discharge/30-day, 12, 24, 36, and 60 months
  Rate of patients with increasing (>5 mm) or stable true lumen in the stented region
Size of false lumen | prior to discharge/30-day, 12, 24, 36, and 60 months
  Rate of patients with stable or decreasing (<5 mm) false lumen in the stented region
Status of false lumen | prior to discharge/30-day, 12, 24, 36, and 60 months
  Rate of patients with obliterated, completely thrombosed, partially thrombosed, or patent false lumen in the stented region (top, middle, 2 cm proximal to distal end), between the bottom of the stent and the celiac trunk, and between the celiac trunk and the aortic bifurcation
Primary entry tear | prior to discharge/30-day, 12, 24, 36, and 60 months
  Rate of patients with covered primary entry tear
Secondary intervention(s) | 30-day, 12, 24, 36, and 60 months
  Rate of patients with secondary intervention(s)
Reintervention(s) | 30-day, 12, 24, 36, and 60 months
  Rate of patients with reintervention(s)
Cerebrovascular event | 30-day, 12, 24, 36, and 60 months
  Rate of patients with new cerebrovascular event/stroke (excluding transient ischemic attack)
Permanent paraplegia | 30-day, 12, 24, 36, and 60 months
  Rate of patients with a new permanent paraplegia
Permanent paraparesis | 30-day, 12, 24, 36, and 60 months
  Rate of patients with a new permanent paraparesis
Migration | prior to discharge/30-day, 12, 24, 36, and 60 months
  Rate of E-nya stent graft migration
  * Rate of patients with proximal E-nya Thoracic Stent Graft migration >5 mm
  * Rate of patients with distal E-nya Thoracic Stent Graft migration >5 mm
Dislodgement | prior to discharge/30-day, 12, 24, 36, and 60 months
  Rate of patients with E-nya Stent Graft dislodgement (full component separation)
Integrity | prior to discharge/30-day, 12, 24, 36, and 60 months
  Rate of patients with failure of E-nya Stent Graft integrity (stent fracture, fabric erosion)
Infolding | prior to discharge/30-day, 12, 24, 36, and 60 months
  Rate of patients with infolding of an E-nya Stent Graft

CONTACTS AND LOCATIONS:
Overall Officials: Jan Brunkwall, Prof., Study Director — Brumed; Jost P. Schäfer, Prof., Study Chair — University Hospital Schleswig-Holstein (UKSH) Kiel
Locations (1):
- Universitätsklinikum Münster, Münster, North Rhine-Westphalia, Germany